CLINICAL TRIAL: NCT07079098
Title: Pilot/Phase I Trial of Oligometastasis SBRT With Immediate, Simulation-Free Treatment Delivery (OLIGO-SWIFT)
Brief Title: Trial of Oligometastasis SBRT With Immediate, Simulation-Free Treatment Delivery (OLIGO-SWIFT)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2Y25
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Oligometastasis; Oligometastatic Disease
Keywords: Stereotactic Body Radiation Therapy; SBRT

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulation-free treatment delivery of SBRT (Experimental)
  Interventions: Other: Simulation-free workflow; Radiation: SBRT

INTERVENTIONS:
Other: Simulation-free workflow — Pre-existing diagnostic images (CTs, PET/CTs, or MRIs) will be imported into the online treatment planning system called Ethos. The Ethos platform and online adaptive radiation therapy (ART) will be utilized at the time of treatment planning and the first (of five) fractions. Subsequent fractions will be delivered using standard image-guided radiotherapy (IGRT) or ART; this will be decided by the treating physician and institutional guidelines.
Radiation: SBRT — Participants will receive SBRT per standard of care in up to five fractions. Fractions will be delivered once daily or once every other day over a total period of one to two weeks.

SUMMARY:
This study is for participants whose cancer is oligometastatic, meaning it has spread to up to five spots in their body and their doctor recommends that they have stereotactic body radiation therapy (SBRT) to treat these cancer sites. SBRT is a type of radiation therapy that may help people with oligometastatic disease live longer without cancer progression. SBRT is usually given in addition to other cancer treatments, like chemotherapy, immunotherapy, or hormone therapy.

Preparing for SBRT can take up to a week or longer. This can make it harder for participants to receive SBRT and coordinate care. This can also mean a longer time until symptoms from cancer sites improve. Doctors would like to treat oligometastatic cancers more quickly by reducing the time it takes to plan for the SBRT.

The typical workflow for SBRT includes doctors doing a simulation which requires a CT (Computerized Tomography) scan. The CT scan is used to create a treatment plan. It can take time to schedule this CT scan and then it normally takes another 5-10 days to create a treatment plan.

A way to reduce the planning time for SBRT is to use the CT scan (or other radiology scan types, like magnetic resonance imaging [MRI] or positron emission tomography [PET]) that participants had when their cancer was diagnosed to plan their SBRT. This eliminates the scheduling of an additional CT scan and the 5-10 day planning time. This is called CTsim-free (CT simulation-free) treatment planning.

CT-sim-free radiation therapy planning has been shown to be effective in treating cancers that are causing pain in people with more advanced or widespread cancers. This study is being done to find out if it is safe and effective to use CTsim-free planning for SBRT to treat oligometastases.

DETAILED DESCRIPTION:
Oligometastatic disease (OMD) is a clinical evolution of cancer in which it has spread beyond the primary site but is not yet broadly metastatic. Oligometastases in radiation oncology are typically defined as being 1 to 5 metastatic lesions that can be safely treated with or without a controlled primary tumor. While multiple factors, including individual's overall health, tumor characteristics and treatment goals, play a crucial role in determining the most appropriate multidisciplinary approach to treating OMD, stereotactic body radiation therapy (SBRT) remains a cornerstone in the standard of care for local OMD therapy and data from multiple clinical trials conducted over several years proved its efficacy in the treatment of oligometastases.

However, traditional SBRT plan generation is a time-consuming process that involves thorough effort. A plan can take up to 5 to 10 working days to be generated in addition to CT-simulation as well as multiple clinical and treatment visits. As the time factor is essential in radiation oncology (RO), extended time to delivery can be a strain for people with OMD. This is particularly challenging in OMD due to the multiple disease sites for treatment (up to 5 in a course) as well as the need to coordinate care with ongoing systemic therapy, which often requires safety washout windows around SBRT, but for which prolonged treatment gaps are often undesirable for systemic control. In an attempt to expedite the time-consuming and lengthy overall treatment time, as well as the potential benefit for people with OMD to receive quick treatment a better optimized workflow is needed.

A proposed solution for expedited SBRT for OMD is the use of simulation-free radiation treatment planning, in which pre-existing diagnostic images are used to generate a radiation treatment pre-plan (as opposed to acquiring planning-specific image sets). This can be implemented using with online adaptive radiotherapy (ART) to refine and finalize the treatment plan at the time of first-fraction delivery, rather than using a standard simulation process. To account for inconsistencies between diagnostic CT and treatment sessions, automated treatment planning is critical for providing rapid online adaptive radiation therapy with full re-optimization based on the anatomy of the day. This can speed up the process of treatment delivery and optimize on-table dose computation. ART has been proven as clinically feasible and time-efficient in prospective clinical trials treating other anatomical sites. Similarly, simulation-free treatment is an emerging standard of care for urgent, palliative radiotherapy settings. However, to date, the feasibility of simulation-free SBRT using an online ART workflow for oligometastases has not been prospectively tested.

Therefore, the purpose of this study is to demonstrate the feasibility of a simulation-free workflow for oligometastases SBRT using online ART. 15 participants will be enrolled; 5 participants with treatment sites in the thorax, 5 with treatment sites in the abdomen/pelvis, and 5 with treatment sites in non-spine bone.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically, cytologically, or radiographically or confirmed cancer that is oligometastastatic (defined in this protocol as up to 5 active sites of disease at time of trial enrollment). Note that previous ablative therapy to the treatment site (excluding prior external beam radiation) is permitted, such as previous microwave ablation or radiofrequency ablation.
* Age ≥18 years.
* Performance status: Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2
* Estimated life expectancy of at least 3 months
* Participants must be considered a candidate for SBRT by the treating physician
* Prior chemotherapy or biological treatment is allowed, but any active oncological treatment should be stopped at least 1 week prior to radiation therapy and renewed no sooner than 1 week following radiation therapy, with the exception of endocrine therapies, which can continue through radiation treatment.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.
* Participants must have a diagnostic CT, MRI, or PET/CT of the site(s) intended for treatment, with or without contrast, acquired no more than 30 days prior to study consent.

Exclusion Criteria:

* Prior radiotherapy to any site overlapping with the projected site for protocol treatment.
* Participants with isolated vertebral metastases except for sacral spine; participants with osseous spine disease can be treated upon this protocol, but those sites (cervical, thoracic, lumbar spine) are not permitted for treatment upon this study. Such participants could be enrolled for treatment to other, concurrent (e.g., visceral, or non-spine bone) disease on this study.
* Pregnant or breastfeeding women are excluded from this study.
* Women of childbearing potential must have a negative pregnancy test within 14 days of study entry. If pregnancy test is not clinically indicated as determined by the treating physician or protocol principal investigator (PI), documentation of this exception is sufficient in lieu of a pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a simulation-free adaptive radiotherapy approach for oligometastasis SBRT in clinical settings, as measured by successful completion of treatment | Up to 2 weeks (timeframe of SBRT treatment)
  Successful completion of treatment will be determined by first-fraction radiation delivery occurring in the first on-table treatment attempt for at least 70% of participants with simulation-free plans meeting dosimetric requirements.
Feasibility of a simulation-free adaptive radiotherapy approach for oligometastasis SBRT in clinical settings, as measured by pre-treatment quality assurance clinical gamma passing index | Up to 2 weeks (timeframe of SBRT treatment)
  A pre-treatment quality assurance clinical gamma passing index that is less than or equal to 2%/2mm will be considered successful.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Henke, MD, MSCI, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No